CLINICAL TRIAL: NCT02942134
Title: Acquisition and Evaluation of Augemented Dyspnea After Use of Non-invasive Ventilation in Patients With COPD and Empysema (Deventilation Syndrome)
Brief Title: Acute Dyspnea After Use of Non-invasive Ventilation in COPD and Emphysema (Deventilation Syndrome)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Felix JF Herth (Other)
Responsible Party: Sponsor-Investigator, Felix JF Herth, Prof. Dr. med. Felix JF Herth, Heidelberg University
Organization: Heidelberg University (Other)
Other Study IDs: S-484/2016
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Obstructive Chronic Bronchitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute dyspnea after use of non-invasive ventilation (NIV) is a common phenomenon in patients with COPD and emphysema. This trial aims to document incidence and severity of augmented dyspnea in patients with long term NIV therapy. These findings may help in understanding the pathomechanisms that lead to post-NIV dyspnea and thus give way to potential therapy schemes.

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) is a widespread therapy option for patients with hypercapnic failure due to COPD and emphysema. Augmented dyspnea after use of NIV is commonly found and leads not only to high patient discomfort, but can also be associated with acute respiratory failure. This monocentric obervation trial includes patients with COPD III°-IV° (GOLD) and emphysema and an established long term NIV therapy. During their routine inpatient follow-up, we will extend the routine examinations, focussing on the vulnerable first hour after the nocturnal use of NIV. This includes monitoring of breath rate, heart rate, pulsoxymetry, trancutaneous CO2, blood pressure and capillary blood gas analysis. Sonographic measurement of diaphragm movement and thickness will be complemented. Subjective dyspnea will be documented by use of the BORG scale.

By collecting this data, we hope to understand the pathomechanisms causing augmented dyspnea after NIV and thus provide information for therapeutical concepts to prevent it.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with stabile COPD, last exacerbation over one month,
* GOLD III to IV
* Regular use of noninvasive ventilation, more than four hours per day for more than one year
* Signed declaration of consent
* Sufficient language capabilities, german

Exclusion Criteria:

* Acute exacerbation in the past four weeks
* Acute pulmonary embolus
* Haemoptysis
* Severe neurological disease
* Severe cardiological disease
* Haemodynamic instability
* New hypoxia or worsening of hypercapnia more than twenty percent of usual rate
* Acute pneumothorax
* Other instable Situation, for example intraabdominal bleedings
* Drug or alcohol dependency
* Regular intake of morphium
* Adiposity BMI over 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hypercapnic failure due to COPD III to IV GOLD and emphysema on long term noninvasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of acute dyspnea after use of non-invasive Ventilation in COPD and emphysema | May 2018

CONTACTS AND LOCATIONS:
Overall Officials: Felix FJ Herth, Prof., Principal Investigator — Medical Director Thoraxklinik Heidelberg

IPD SHARING:
Plan to Share IPD: No